CLINICAL TRIAL: NCT01605266
Title: INSIGHT (Insight Into Nephrotic Syndrome: Investigating Genes, Health and Therapeutics)
Brief Title: INSIGHT (Insight Into Nephrotic Syndrome)
Acronym: INSIGHT
Status: Recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Rulan Parekh, Staff Physician, The Hospital for Sick Children
Other Study IDs: 1000021384
Record Dates: First submitted 2012-04-20; First posted 2012-05-24 (Estimated); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Nephrotic Syndrome
Keywords: pediatric; kidney disease; minimal change disease; focal segmental glomerulosclerosis; nephrotic syndrome
MeSH Terms: conditions — Nephrotic Syndrome; Kidney Diseases; Nephrosis, Lipoid; Glomerulosclerosis, Focal Segmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood is drawn for DNA, serum, plasma, buffy coat and whole blood. Urine and toenail clippings are also collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nephrotic Syndrome: The cohort includes all children diagnosed with nephrotic syndrome between ages 1-18. Children and their caregiver must be willing to provide informed consent, complete questionnaires, and provide biospecimens of the child. Those with secondary causes of nephrotic syndrome and/or systemic disease are excluded.

SUMMARY:
INSIGHT is a longitudinal study of childhood nephrotic syndrome to determine genetic, serologic and environmental factors contributing to nephrotic syndrome and disease progression.

DETAILED DESCRIPTION:
INSIGHT is a longitudinal observational study of childhood nephrotic syndrome to determine genetic, serologic and environmental factors contributing to nephrotic syndrome and disease progression. This is a large multiethnic cohort to test hypotheses of gene and environmental risk factors and disease progression. Participants are recruited from Toronto, Ontario and surrounding regions. Additional sites will be added on in the future.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of nephrotic syndrome
2. signed informed consent and assent appropriate for age
3. ages 6 months -18 years old and
4. ability to complete questionnaires

Exclusion Criteria:

1. congenital nephrotic syndrome (less than age 1)
2. syndromic disease with multiple organ involvement
3. inability to provide consent by primary care providers
4. conditions such as systemic lupus erythematous.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with nephrotic syndrome. Children are recruited from Toronto and surrounding region with additional sites added later.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-01; Primary Completion 2032-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Relapse (number of relapses) | Entire follow-up
  After remission, an increase in the first AM morning urine protein ≥ 3+ for 3 consecutive days or increase in maintenance prednisone dose

SECONDARY OUTCOMES:
Frequently relapsing NS (yes or no) | 6, 12, 18 and 24 months
  4 or more relapses within any 12 month interval OR 2 or more relapses within the first 6 months since diagnosis
Steroid - dependent NS (yes or no) | 6, 12, 18 and 24 months
  2 relapses during steroid taper or a relapse within 14 days of steroid discontinuation
Initial Steroid Resistance (yes or no) | Up to 16 weeks
  Commencing second line medication due to no response from prednisone with initial treatment
CKD (yes or no) | Entire follow-up
  eGFR less than or equal to 60mg/ml/1.73m^2 for 3 or more consecutive months
ESRD (yes or no) | Entire follow-up
  eGFR less than or equal to 15 mg/ml/1.73m^2, or initiation of dialysis or receiving a transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Rulan Parekh, MD, Principal Investigator — The Hospital for Sick Children
Locations (4):
- Canada (4):
  - William Osler Health System, Brampton Civic Hospital and Peel Memorial Centre for Integrated Health and Wellness, Brampton, Ontario
  - Hamilton Health Sciences Corporation - McMaster University Medical Centre, Hamilton, Ontario
  - Rouge Valley Health System, Rouge Valley Centenary, Scarborough Village, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hussain N, Zello JA, Vasilevska-Ristovska J, Banh TM, Patel VP, Patel P, Battiston CD, Hebert D, Licht CP, Piscione TD, Parekh RS. The rationale and design of Insight into Nephrotic Syndrome: Investigating Genes, Health and Therapeutics (INSIGHT): a prospective cohort study of childhood nephrotic syndrome. BMC Nephrol. 2013 Jan 26;14:25. doi: 10.1186/1471-2369-14-25. PMID 23351121
- [Result] Borges K, Vasilevska-Ristovska J, Hussain-Shamsy N, Patel V, Banh T, Hebert D, Pearl RJ, Radhakrishnan S, Piscione TD, Licht CP, Langlois V, Levin L, Strug L, Parekh RS. Parental attitudes to genetic testing differ by ethnicity and immigration in childhood nephrotic syndrome: a cross-sectional study. Can J Kidney Health Dis. 2016 Mar 17;3:16. doi: 10.1186/s40697-016-0104-y. eCollection 2016. PMID 26998310
- [Result] Banh THM, Hussain-Shamsy N, Patel V, Vasilevska-Ristovska J, Borges K, Sibbald C, Lipszyc D, Brooke J, Geary D, Langlois V, Reddon M, Pearl R, Levin L, Piekut M, Licht CPB, Radhakrishnan S, Aitken-Menezes K, Harvey E, Hebert D, Piscione TD, Parekh RS. Ethnic Differences in Incidence and Outcomes of Childhood Nephrotic Syndrome. Clin J Am Soc Nephrol. 2016 Oct 7;11(10):1760-1768. doi: 10.2215/CJN.00380116. Epub 2016 Jul 21. PMID 27445165
- [Result] Borges K, Sibbald C, Hussain-Shamsy N, Vasilevska-Ristovska J, Banh T, Patel V, Brooke J, Piekut M, Reddon M, Aitken-Menezes K, McNaughton A, Pearl RJ, Langlois V, Radhakrishnan S, Licht CPB, Piscione TD, Levin L, Noone D, Hebert D, Parekh RS. Parental Health Literacy and Outcomes of Childhood Nephrotic Syndrome. Pediatrics. 2017 Mar;139(3):e20161961. doi: 10.1542/peds.2016-1961. Epub 2017 Feb 17. PMID 28213606
- [Result] Konstantelos N, Banh T, Patel V, Vasilevska-Ristovska J, Borges K, Hussain-Shamsy N, Noone D, Hebert D, Radhakrishnan S, Licht CPB, Langlois V, Pearl RJ, Parekh RS. Association of low birth weight and prematurity with clinical outcomes of childhood nephrotic syndrome: a prospective cohort study. Pediatr Nephrol. 2019 Sep;34(9):1599-1605. doi: 10.1007/s00467-019-04255-1. Epub 2019 Apr 11. PMID 30976899
- [Result] Riar SS, Banh THM, Borges K, Subbarao P, Patel V, Vasilevska-Ristovska J, Chanchlani R, Hussain-Shamsy N, Noone D, Hebert D, Licht CPB, Langlois V, Pearl RJ, Parekh RS. Prevalence of Asthma and Allergies and Risk of Relapse in Childhood Nephrotic Syndrome: Insight into Nephrotic Syndrome Cohort. J Pediatr. 2019 May;208:251-257.e1. doi: 10.1016/j.jpeds.2018.12.048. Epub 2019 Feb 4. PMID 30732999
- [Derived] Robinson CH, Aman N, Banh THM, Brooke J, Dhillon V, Garner M, Licht C, McKay A, Pearl R, Radhakrishnan S, Rasool K, Selvathesan N, Teoh CW, Vasilevska-Ristovska J, Parekh RS. Challenging Clinical Practice Guideline Definitions in Childhood Nephrotic Syndrome. Clin J Am Soc Nephrol. 2025 Dec 1;20(12):1767-1779. doi: 10.2215/CJN.0000000842. Epub 2025 Oct 15. PMID 41091558
- See also: PubMed: The rationale and design of Insight into Nephrotic Syndrome: Investigating Genes, Health and Therapeutics (INSIGHT): a prospective cohort study of childhood nephrotic syndrome. — http://www.ncbi.nlm.nih.gov/pubmed/23351121